CLINICAL TRIAL: NCT04120870
Title: Comparison of Effects on Hemodynamics Between Ketamine and Etomidate During Rapid Sequence Intubation in Trauma Patients With High Shock Index
Brief Title: Comparison of Ketamine and Etomidate During Rapid Sequence Intubation in Trauma Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulties in obtaining consent because of emergency situation
Sponsor: Ajou University School of Medicine (Other)
Collaborators: Unimedics (http://unimedics.co.kr) (Unknown)
Responsible Party: Principal Investigator, In-kyong Yi, Clinical assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MED-OBS-19-294
Record Dates: First submitted 2019-09-26; First posted 2019-10-09 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Trauma; Shock, Traumatic
Keywords: etomidate; ketamine; rapid sequence intubation; trauma; hemodynamics
MeSH Terms: conditions — Wounds and Injuries; Shock, Traumatic | interventions — Etomidate; Ketamine

STUDY DESIGN:
Intervention Model Description: ketamine group: ketamine 2 mg/kg iv as induction agent etomidate group: etomidate 0.2 mg/kg iv as induction agent
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etomidate (Active Comparator): The induction agent of rapid sequence intubation is etomidate. 0.2 mg/kg
  Interventions: Drug: Etomidate Injection 0.2 mg/kg
- Ketamine (Experimental): The induction agent of rapid sequence intubation is ketamine. 2 mg/kg
  Interventions: Drug: Ketamine injection 2 mg/kg

INTERVENTIONS:
Drug: Etomidate Injection 0.2 mg/kg — The induction agent of rapid sequence intubation is etomidate. 0.2 mg/kg
  Other Names: Etomidate
  Arms: Etomidate
Drug: Ketamine injection 2 mg/kg — The induction agent of rapid sequence intubation is ketamine. 2 mg/kg
  Other Names: Ketamine
  Arms: Ketamine

SUMMARY:
In trauma patients with high shock index, the investigators compare the effects on hemodynamics between ketamine and etomidate.

DETAILED DESCRIPTION:
In trauma patients, rapid sequence intubation is recommended. The drug of choice, however, has been debated. One cohort comparative study showed ketamine had benefit in hemodynamics compared to etomidate in trauma patients. One observational study showed in high shock index patients, ketamine showed maintain systolic blood pressure. And other retrospective showed less clinical hypotension was less in ketamine. However there is no randomized controlled study comparing ketamine and etomidate in trauma patients. The purpose of this study is comparing the effects of hemodynamics between ketamine and etomidate in high shock index trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* age 19~70
* Shock index ≥ 0.9
* Patients who need intubation regarding to Ajou trauma center protocol

Exclusion Criteria:

* during CPR
* CPR before hospital arrival
* Severe head trauma
* Steroid intake history

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure difference compared with baseline after 10 minutes | 13 minutes
  Systolic blood pressure 10 minutes after induction agent injection - baseline systolic blood pressure mmHg Positive or zero value means good result. Negative value means poor result.

SECONDARY OUTCOMES:
Intubating condition | 5 minutes
  Intubator judge intubating condition Laryngoscopy: easy / fair / difficult (difficult is the worst result) Vocal cords position: abducted / moving / closed (closed is the worst result) Reaction to insertion of the tracheal tube and cuff inflation : none / slight / vigorous (none is the worst result)
  If one of category checked the worst score, it considered :clinically unacceptable".
Incidence of hypotension | 25 minutes
  If any of these are checked, define as hypotension (from injection of induction agent to 20 minutes after)
  1. systolic pressure < 90 mmHg
  2. systolic pressure decrease > 40% compared to baseline
  3. Initiation of vasopressor
  4. Vasopressor dose increase > 30% of initial vaopressor dose
  5. Fluid or blood loading
  Patient numbers (%)
Incidence of hypertension | 25 miinutes
  From injection of induction agent to 20 minutes after, systolic pressure > 160 mmHg defined as hypertension
  Patients numbers (%)

CONTACTS AND LOCATIONS:
Overall Officials: In Kyong Yi, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou university school of medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
If there is a reasonable request, we can share the data personally.